CLINICAL TRIAL: NCT06301191
Title: The Effect of Semaglutide on Endothelial Function, Arterial Stiffness and Liver Indices in Patients Witn Type 2 Diabetes Mellitus and NAFLD
Brief Title: The Effect of Semaglutide on Cardiovascular Markers and Liver Function
Status: Recruiting | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Professor of Internal Medicine-Endocrinology, Attikon Hospital
Other Study IDs: 133/21-02-2022
Record Dates: First submitted 2024-02-29; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Blood sample obtained from the subjects for oxidative stress markers (malondialdehyde and protein carbonyls), nitrites and nitrates, N-terminal pro B-type natriuretic peptide (NT-proBNP) measuring.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Semaglutide group: 25 patients treated with semaglutide. Pulse wave velocity, aumentation index, SBPao and PPao with Arteriograph, Mobilograph and Complior, and perfused boundary region (PBR) of sublingual vessels using a high-resolution camera with Sideview Darkfield Imaging technique (Microscan, Glucockeck) will be evaluated. PBR consists the cell-free space which is formed from the separation of red blood cells from plasma at the surface of the endothelial glycocalyx.Liver steatosis and stiffness will be measured using Fibroscan® Mini+ 430 (Echosens, Paris, Île-de-France). CAP score will be used as an index of liver fat content, with normal values being < 238 dB/m. E score will be used as an index of liver fibrosis, with normal values being 2- 6 kPa. Blood glucose, glycosylated hemoglobin (HbA1c) and a full lipidemic profile will be measured before and at 4 and 12 months of treatment.
  Interventions: Drug: Semaglutide, 1.0 mg/mL
- D-PP4 group: 25 patients treated with D-PP4 inhibitors. Pulse wave velocity, augmentation index, SBPao and PPao with Arteriograph, Mobilograph and Complior, and perfused boundary region (PBR) of sublingual vessels using a high-resolution camera with Sideview Darkfield Imaging technique (Microscan, Glucockeck) will be evaluated. PBR consists the cell-free space which is formed from the separation of red blood cells from plasma at the surface of the endothelial glycocalyx.Liver steatosis and stiffness will be measured using Fibroscan® Mini+ 430 (Echosens, Paris, Île-de-France). CAP score will be used as an index of liver fat content, with normal values being < 238 dB/m. E score will be used as an index of liver fibrosis, with normal values being 2- 6 kPa. Blood glucose, glycosylated hemoglobin (HbA1c) and a full lipidemic profile will be measured before and at 4 and 12 months of treatment
  Interventions: Drug: Dipeptidyl Peptidase 4 inhibitor

INTERVENTIONS:
Drug: Semaglutide, 1.0 mg/mL — Semaglutide, 1.0 mg/mL
  Groups: Semaglutide group
Drug: Dipeptidyl Peptidase 4 inhibitor — Dipeptidyl Peptidase 4 inhibitor
  Groups: D-PP4 group

SUMMARY:
Fifty patients with diabetes mellitus type 2 and non-alcoholic fatty liver disease (NAFLD) will be enrolled in the study.

25 patients will treated with semaglutide and 25 patients with dipeptidyl peptidase 4 (D-PP4) inhibitors.

At baseline, at four and at 12 months will evaluate the endothelial, cardiovascular and liver function.

DETAILED DESCRIPTION:
The cardiovascular benefits of semaglutide are established; however, its effect on surrogate vascular markers and liver function is not known.The aim of our study is to investigate the effects of semaglutide on vascular,endothelial and liver function in patients with type 2 diabetes and non-alcoholic fatty liver disease.

A.Overall, 50 patients with diabetes mellitus type 2 and NAFLD will be studied at baseline ,at four and twelve months of treatment:

25 patients will be treated with semaglutide 25 patients will be treated with D-PP4 inhibitors. B. In all patients, the investigators will measure the pulse wave velocity (measured in m/s), pulse wave augmentation index [which is calculated by the formula (P2-P1)/PP x 100, where P1 stands for peak systolic pressure, P2 stands for second peak systolic pressure due to wave reflection and PP stands for Pulse Pressure ], central systolic blood pressure (SBPao, measured in mm Hg) and central pulse pressure (PPao, measured ) with Arteriograph, Mobilograph and Complior, and perfused boundary region of sublingual vessels (5-25 μm in size) using a high-resolution camera with Sideview Darkfield Imaging technique (Microscan, Glucockeck). Perfused boundary region consists the cell-free space which is formed from the separation of red blood cells from plasma at the surface of the endothelial glycocalyx. Increased Perfused boundary region is considered to be an accurate indicator of the reduction of endothelial glycocalyx thickness due to plasma penetration into the glycocalyx.Liver steatosis and stiffness will be measured using Fibroscan® Mini+ 430 (Echosens, Paris, Île-de-France). Controlled Attenuation Parameter (CAP) score will be used as an index of liver fat content, with normal values being < 238 dB/m. E score will be used as an index of liver fibrosis, with normal values being 2- 6 kPa.

The examination will be carried out at the Laboratory of Preventive Cardiology of the 2nd Department of Cardiology of the University of Athens at "Attikon" Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus type 2
* NAFLD

Exclusion Criteria:

* malignancies
* chronic inflammatory disease
* chronic kidney disease (estimated glomerular filtration rate <60 ml/min/m2 for a period of at least 90 days)
* peripheral vascular disease
* retinopathy
* previous therapy with a Glucagon-like peptide-1 agonist.
* None of the female patients was on hormone replacement treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 subjects with T2DM and NAFLD, who attended the Diabetes Outpatients Clinic were enrolled in the study. 25 patients will reciece semaglutide 1 mg (treatment group) and 25 patients will receive DPP-4 inhibitors (either linagliptin or alogliptin or vildagliptin or sitagliptin - control group). Exclusion criteria were malignancies, chronic inflammatory disease, chronic kidney disease (estimated glomerular filtration rate <60 ml/min/m2 for a period of at least 90 days) peripheral vascular disease, retinopathy, and previous therapy with a Glucagon-like peptide-1 agonist. None of the female patients was on hormone replacement treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of arterial stiffness markers difference among treatment groups | 12 months
  Comparison of pulse wave velocity difference among treatment groups. Two non-invasive pressure sensors will be used to record the carotid and femoral waveforms and the distance between the two arterial sites will be measured with a tape measure. Pulse wave velocity is calculated as the distance divided by transit time between waves (m/s).
Comparison of endothelial glycocalyx thickness difference among treatment groups | 12 months
  The investigators will measure the perfused boundary region (PBR) of the sublingual arterial microvessels (ranged from 5 to 25 μm) using Sidestream Darkfield imaging that provides a direct, noninvasive, and fast method for the assessment of the endothelial glycocalyx. The PBR is the cell-poor layer which results from the phase separation between the flowing red blood cells (RBC) and plasma on the surface of the microvessel lumen. The PBR includes the most luminal part of glycocalyx that does allow cell penetration. Thus, an increased perfused boundary region is consistent with deeper penetration of erythrocytes into glycocalyx, indicating a loss of glycocalyx barrier properties and is a marker of reduced glycocalyx thickness.
Comparison of liver stiffness difference among treatment groups | 12 months
  CAP score will be used as an index of liver fat content, with normal values being < 238 dB/m. <237 dB/m (S0, no steatosis), 237 -259 dB/m (S1, mild steatosis), 259 -291 dB/m (S2, moderate steatosis), and 291 -400 dB/m (S3,severe steatosis). E score will be used as an index of liver fibrosis. The cut-off values for fibrosis (F) were as follows:(1) <5.5 kPa (F0, no fibrosis), (2) 5.5-8.0 kPa (F1, mild fibrosis), (3) 8.0-10.0 kPa (F2, moderate fibrosis),(4) 11.0-16.0 kPa (F3, severe fibrosis), and (5) >16.0 kPa (F4, cirrhosis).

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon University General Hospital, Athens, Greece